CLINICAL TRIAL: NCT05752422
Title: Transcranial Photobiomodulation for Adult ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CNS Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNS11082019
Record Dates: First submitted 2019-11-11; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: ADHD
Keywords: ADHD; Attention; Photobiomodulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial Photobiomodulation (t-PBM) (Experimental): Active t-PBM will be delivered to the forehead using the Niraxx Smart Headband (gen 1). Daily treatments of 40 min
  Interventions: Device: Niraxx G1 Headband Device including sham
- Sham t-PBM (Sham Comparator): To the subjects belonging to the sham arm the sham treatment sessions will be performed using the same device, during the same time but the device will not be turned on.
  Interventions: Device: Niraxx G1 Headband Device including sham

INTERVENTIONS:
Device: Niraxx G1 Headband Device including sham — Exploring effect of active t-PBM delivered by Niraxx G1 Headband versus sham condition

SUMMARY:
This study aims to assess the behavioral as well cognitive changes in ADHD symptoms in terms of improvement of inhibitory control and attention in adults with ADHD

DETAILED DESCRIPTION:
This study is a randomized double blind trial. After selection and enrollment, participants will be screened at baseline with a complete diagnostic and clinical assessment, and randomized to receive active or placebo t-PBM.

At visit 1 patients will undergo a (pre-treatment) neuropsychological testing followed by the first t-PBM session. After the first t-PBM session, the patients will undergo another (post-treatment) neuropsychological testing. After visit 1, which includes the first treatment, patients will receive additional 4 weeks of t-PBM treatments. After the last treatment, patients will come to clinic for undergo a clinical and neuropsychological assessment (visit 2). After the visit 2, patients will receive other 4 weeks of t-PBM treatments. After the last t-PBM treatment session, patients will come to clinic to undergo the final clinical and neuropsychological assessment (visit 3).

At the visits 1, 2 and 3 patients will be asked if they believe they received active or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

• subjects diagnosed with ADHD

Exclusion Criteria:

* schizophrenia or other psychosis
* current acute depressive episode
* bipolar disorder with current manic or depressive episode
* active substance use disorder
* autism
* dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
4-weeks effect of t-PBM | 1 month
  To assess the effects of 4 weeks PBM treatment in terms of improvement of inhibitory control, as assessed through the Stop Signal Task
4-weeks effect of t-PBM | 1 month
  To assess the cognitive changes of 4 weeks PBM treatment in terms of improvement of normalization of intra-individual reaction time variability as assessed through the Stop Signal Task
4-weeks effect of t-PBM | 1 month
  To assess the clinical changes of 4 weeks PBM treatment in terms of reduction of ADHD symptoms severity
8-weeks effect of t-PBM | 2 months
  To assess the behavioral/cognitive and clinical changes of 8 weeks PBM treatment in terms of improvement of inhibitory control and normalization of intra-individual reaction time variability, as assessed through the Stop Signal Task, as well reduction of ADHD symptoms severity
8-weeks effect of t-PBM | 2 months
  To assess the behavioral changes of 8 weeks PBM treatment in terms of improvement of inhibitory control, as assessed through the Stop Signal Task
8-weeks effect of t-PBM | 2 months
  To assess the cognitive changes of 8 weeks PBM treatment in terms of normalization of intra-individual reaction time variability, as assessed through the Stop Signal Task
8-weeks effect of t-PBM | 2 months
  To assess the clinical changes of 8 weeks PBM treatment in terms of reduction of ADHD symptoms severity

REFERENCES:
- [Background] American Psychiatric Association, 2013. Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Diagnostic Stat. Man. Ment. Disord. 4th Ed. TR. 280. Caldieraro, M. A., & Cassano, P. (2019). Journal of Affective Disorders Transcranial and systemic photobiomodulation for major depressive disorder : A systematic review of efficacy , tolerability and biological mechanisms. Journal of Affective Disorders, 243(May 2018), 262-273. https://doi.org/10.1016/j.jad.2018.09.048 Hwang, J, Castelli, D. M, Gonzalez-Lima, F, 2016. Cognitive enhancement by transcranial laser stimulation and acute aerobic exercise. Lasers in Medical Science 31-6, 1151-1160 Barrett, D. W. (2013). Transcranial Infrared Laser Stimulation Produces Beneficial Cognitive And Emotional Effects In Humans. Neuroscience, 230, 13-23. https://doi.org/10.1016/j.neuroscience.2012.11.016